CLINICAL TRIAL: NCT04844944
Title: The Helios Heart Registry: A Standardized Registry for Capturing Clinical and Patient-reported Outcomes in Patients With Specific Cardiac Diseases: Application of the ICHOM Standard in Clinical Practice
Brief Title: The Helios Heart Registry: A Standardized Registry for Patients With Specific Cardiac Diseases
Acronym: H²-Registry
Status: Recruiting | Type: Observational
Sponsor: Helios Health Institute GmbH (Other)
Responsible Party: Sponsor
Other Study IDs: 2021-0016
Record Dates: First submitted 2021-03-29; First posted 2021-04-14 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-10

CONDITIONS: Heart Failure; Coronary Artery Disease; Atrial Fibrillation
Keywords: cardiovascular disease; HF; CAD; AF; ICHOM
MeSH Terms: conditions — Heart Failure; Coronary Artery Disease; Atrial Fibrillation; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Heart Failure: Hospitalized patients diagnosed with Heart Failure. No Intervention.
- Coronary Artery Disease: Hospitalized patients diagnosed with Coronary Artery Disease. No Intervention.
- Atrial Fibrillation: Hospitalized patients diagnosed with Atrial Fibrillation. No Intervention.

SUMMARY:
Investigator-initiated, prospective, non-randomized, open label, non-interventional multicenter registry to evaluate current treatment of three major cardiovascular disease entities in clinical practice using a standardized variable-set of relevant covariates and outcome measures.

DETAILED DESCRIPTION:
Heart failure (HF), coronary artery disease (CAD) and atrial fibrillation (AF) are among the most relevant cardiovascular diseases contributing to overall morbidity and mortality each itself and in particular in case of their coexistence. Several new therapies have been introduced in randomized controlled trials but confirmation data of treatment effects in real-world cohorts using a standardized methodology is scarce. The International Consortium for Health Outcomes Measurement (ICHOM) defined standard variable sets for all three diseases in order to objectively monitor the course of disease.

To evaluate current health care utilization and interactions between diseases and treatments in patients with HF, CAD and AF as well as patient-oriented values study initiator will build a prospective, observational, multicenter cardiovascular registry using standardized patient variables and endpoints based on the ICHOM recommendations.

ELIGIBILITY:
Inclusion Criteria:

* Age of 18 years or older
* Inpatient Treatment
* Present diagnosis of at least one of the three cardiovascular disease entities of interest according to the current guidelines of the European Society of Cardiology (ESC): HF, CAD, AF

Exclusion Criteria:

* Inability to provide informed consent
* Initial presentation (index hospitalization) in cardiogenic shock or other kinds of shock
* Patient after heart transplantation or patient with present ventricular assist device (VAD)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients being admitted as inpatients to a cardiology ward of one of the participating centers with one or more major cardiovascular disease entities (HF, CAD, AF)
Sampling Method: Probability Sample
Enrollment: 24000 (Estimated)
Dates: Start 2021-03-30 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
All-cause mortality during f/u | 6 months
All-cause mortality during f/u | 12 months
All-cause mortality during f/u | 18 months

SECONDARY OUTCOMES:
in-hospital mortality | 3 days
cardiovascular mortality during f/u | 6 months
cardiovascular mortality during f/u | 12 months
cardiovascular mortality during f/u | 18 months
length of hospital stay | 3 days
rate of rehospitalizations of any cause during f/u | 6 months
rate of rehospitalizations of any cause during f/u | 12 months
rate of rehospitalizations of any cause during f/u | 18 months
rate of rehospitalizations for cardiovascular causes during f/u | 6 months
rate of rehospitalizations for cardiovascular causes during f/u | 12 months
rate of rehospitalizations for cardiovascular causes during f/u | 18 months
rate of rehospitalizations for specific cardiovascular diseases | 6 months
rate of rehospitalizations for specific cardiovascular diseases | 12 months
rate of rehospitalizations for specific cardiovascular diseases | 18 months
rate of specific cardiovascular events | 6 months
rate of specific cardiovascular events | 12 months
rate of specific cardiovascular events | 18 months
general quality of life (PROMIS) | 6 months
general quality of life (PROMIS) | 12 months
general quality of life (PROMIS) | 18 months
general quality of life (PHQ2) | 6 months
general quality of life (PHQ2) | 12 months
general quality of life (PHQ2) | 18 months
disease specific quality of life (KCCQ-12 [HF]) | 6 months
disease specific quality of life (KCCQ-12 [HF]) | 12 months
disease specific quality of life (KCCQ-12 [HF]) | 18 months
disease specific quality of life (SAQ-7 [CAD]) | 6 months
disease specific quality of life (SAQ-7 [CAD]) | 12 months
disease specific quality of life (SAQ-7 [CAD]) | 18 months
disease specific quality of life (AFEQT [AF]) | 6 months
disease specific quality of life (AFEQT [AF]) | 12 months
disease specific quality of life (AFEQT [AF]) | 18 months
side effects associated with drug treatment | 6 months
  The endpoint will be assessed by trained study personnel by the evaluation of patient interviews and medical records at each FU time point. The outcome is defined as any adverse event or known side effect likely attributed to the heart failure related drug therapy leading to consultation of a medical facility or discontinuation of treatment that became apparent after the last study visit.
side effects associated with drug treatment | 12 months
  The endpoint will be assessed by trained study personnel by the evaluation of patient interviews and medical records at each FU time point. The outcome is defined as any adverse event or known side effect likely attributed to the heart failure related drug therapy leading to consultation of a medical facility or discontinuation of treatment that became apparent after the last study visit.
side effects associated with drug treatment | 18 months
  The endpoint will be assessed by trained study personnel by the evaluation of patient interviews and medical records at each FU time point. The outcome is defined as any adverse event or known side effect likely attributed to the heart failure related drug therapy leading to consultation of a medical facility or discontinuation of treatment that became apparent after the last study visit.
complications associated with therapeutic interventions | 6 months
  The endpoint will be assessed by trained study personnel by the evaluation of patient interviews and medical records at each FU time point. The outcome is defined as any adverse event likely being associated with a heart failure related procedure (coronary revascularization, valve intervention / surgery, cardiac electronic device implantation) leading to prolonged hospital stay / additional therapeutic interventions / unplanned consultation of medical facilities.
complications associated with therapeutic interventions | 12 months
  The endpoint will be assessed by trained study personnel by the evaluation of patient interviews and medical records at each FU time point. The outcome is defined as any adverse event likely being associated with a heart failure related procedure (coronary revascularization, valve intervention / surgery, cardiac electronic device implantation) leading to prolonged hospital stay / additional therapeutic interventions / unplanned consultation of medical facilities.
complications associated with therapeutic interventions | 18 months
  The endpoint will be assessed by trained study personnel by the evaluation of patient interviews and medical records at each FU time point. The outcome is defined as any adverse event likely being associated with a heart failure related procedure (coronary revascularization, valve intervention / surgery, cardiac electronic device implantation) leading to prolonged hospital stay / additional therapeutic interventions / unplanned consultation of medical facilities.
adherence to therapy | 6 months
  The endpoint will be assessed by trained study personnel by the evaluation of patient interviews at each FU time point. The outcome is defined as the accordance of prescribed and actually taken medication (from the last to the actual study visit) and will be presented as a ratio of the number of drug doses taken to the number of drug doses prescribed.
adherence to therapy | 12 months
  The endpoint will be assessed by trained study personnel by the evaluation of patient interviews at each FU time point. The outcome is defined as the accordance of prescribed and actually taken medication (from the last to the actual study visit) and will be presented as a ratio of the number of drug doses taken to the number of drug doses prescribed.
adherence to therapy | 18 months
  The endpoint will be assessed by trained study personnel by the evaluation of patient interviews at each FU time point. The outcome is defined as the accordance of prescribed and actually taken medication (from the last to the actual study visit) and will be presented as a ratio of the number of drug doses taken to the number of drug doses prescribed.
disease associated treatment costs | 6 months
disease associated treatment costs | 12 months
disease associated treatment costs | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Bollmann, MD, PhD, Study Chair — Heart Center at University of Leipzig
Locations (10):
- Germany (10):
  - Helios Klinikum Berlin-Buch, Berlin
  - Helios Klinikum Erfurt, Erfurt
  - Helios Klinikum Gifhorn, Gifhorn
  - Helios Klinikum Hildesheim, Hildesheim
  - Heart Center Leipzig at University of Leipzig, Leipzig
  - Helios Vogtlandklinikum Plauen, Plauen
  - Helios Klinikum Schwerin, Schwerin
  - Helios Klinikum Siegburg, Siegburg
  - Helios Dr. Horst Schmidt Kliniken Wiesbaden, Wiesbaden
  - Helios Universitätsklinikum Wuppertal, Wuppertal

REFERENCES:
- [Derived] Leiner J, Hohenstein S, Konig S, Kwast S, Nitsche A, Seyfarth M, Baberg H, Lauten A, Neuser H, Staudt A, Tebbenjohanns J, Andrie R, Niehaus M, Ferrari MW, Muller M, Schulte N, Bode K, Kuhlen R, Bollmann A. Characteristics and outcomes of patients with heart failure and reduced left ventricular ejection fraction in relation to sodium-glucose cotransporter-2 inhibitor treatment: real-world data from the multicentre H2-registry. Clin Res Cardiol. 2026 Feb 2. doi: 10.1007/s00392-026-02853-2. Online ahead of print. PMID 41627441
- [Derived] Leiner J, Konig S, Nitsche A, Hohenstein S, Nagel J, Seyfarth M, Baberg H, Lauten A, Neuser H, Staudt A, Tebbenjohanns J, Andrie R, Niehaus M, Ferrari MW, Kuhlen R, Bollmann A. A multicentre registry of hospitalized patients with acute and chronic heart failure: Study design of the H2-registry. ESC Heart Fail. 2025 Aug;12(4):3114-3133. doi: 10.1002/ehf2.15266. Epub 2025 Apr 13. PMID 40222816